CLINICAL TRIAL: NCT03236909
Title: Expanded Indications in the Adult Cochlear Implant Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G170111
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-arm (Experimental): Single-arm, repeated-measures study design with all subjects receiving a MED-EL cochlear implant
  Interventions: Device: MED-EL SYNCHRONY/SYNCHRONY PIN Cochlear Implant System

INTERVENTIONS:
Device: MED-EL SYNCHRONY/SYNCHRONY PIN Cochlear Implant System — Subjects will be implanted with the MED-EL SYNCHRONY/SYNCHRONY PIN Cochlear Implant System with +FLEX28 or +FLEXSOFT electrode arrays. Subjects will be fit with the SONNETEAS (ear-level) and/or RONDO (single-unit) external audio processors.
  Other Names: SYNCHRONY +FLEXSOFT; SYNCHRONY +FLEX28

SUMMARY:
The purpose of this investigation is to expand FDA-approved labeling for MED-EL cochlear implants to include adults who have moderate to profound sensorineural hearing loss and obtain limited benefit from appropriately fit hearing aids.

DETAILED DESCRIPTION:
Fifty (50) subjects, 18 years of age and older, will be implanted across the United States and Canada. Subjects with moderate to profound bilateral sensorineural hearing loss will be implanted with the MED-EL SYNCHRONY/SYNCHRONY PIN Cochlear Implant System. .

Limited benefit from amplification is defined by test scores of 60% correct or less in the ear to be implanted (70% or less in the nonimplanted ear) on monosyllabic words in quiet. Subjects will be followed for twelve (12) months post-activation of the SONNETEAS Audio Processor.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older at the time of implantation
* Moderate to profound hearing loss in the low frequencies and severe to profound hearing loss in the high frequencies, bilaterally as defined by: Low-frequency PTA (250, 500, and 1000 Hz) greater than 40 dB High-frequencies not better than 65 dB (3000 Hz - 8000 Hz)
* Sensorineural hearing loss, demonstrated by an air-bone gap of less than or equal to 10dB
* Limited benefit from appropriately fit hearing aids, defined by CNC word score in quiet of 60% or less in the ear to be implanted and 70% or less in the non-implanted ear
* CNC word score in quiet of greater than or equal to 10% in the ear to be implanted
* Evidence of appropriately fit hearing aids as determined by the audiologist
* Bilateral hearing aids should be considered standard of care, except in situations where the audiologist, physician, or potential subject determines that unilateral fit is optimal
* Hearing aid fit should be verified through accepted measures such as functional gain or real-ear verification
* If appropriately fit hearing aids have not been worn within the last year, a 30-day hearing aid trial must be completed prior to enrollment in the study
* Fluent in English
* No radiological contraindications
* Ability to undergo general anesthesia
* Appropriate motivation and expectation levels
* Stated willingness to comply with all study procedures for the duration of the study

Exclusion Criteria:

* Evidence that hearing loss is retrocochlear in origin
* Active middle ear infection
* Skin or scalp condition precluding use of external audio processor- Suspected cognitive impairment or organic brain dysfunction
* History of prior use of a hearing implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - University of Miami, Miami, Florida
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amoodi HA, Mick PT, Shipp DB, Friesen LM, Nedzelski JM, Chen JM, Lin VY. Results with cochlear implantation in adults with speech recognition scores exceeding current criteria. Otol Neurotol. 2012 Jan;33(1):6-12. doi: 10.1097/MAO.0b013e318239e5a1. PMID 22090001
- [Background] Bassim MK, Buss E, Clark MS, Kolln KA, Pillsbury CH, Pillsbury HC 3rd, Buchman CA. MED-EL Combi40+ cochlear implantation in adults. Laryngoscope. 2005 Sep;115(9):1568-73. doi: 10.1097/01.mlg.0000171023.72680.95. PMID 16148696
- [Background] Cox RM, Alexander GC. The abbreviated profile of hearing aid benefit. Ear Hear. 1995 Apr;16(2):176-86. doi: 10.1097/00003446-199504000-00005. PMID 7789669
- [Background] Cullen RD, Higgins C, Buss E, Clark M, Pillsbury HC 3rd, Buchman CA. Cochlear implantation in patients with substantial residual hearing. Laryngoscope. 2004 Dec;114(12):2218-23. doi: 10.1097/01.mlg.0000149462.88327.7f. PMID 15564849
- [Background] Dorman MF, Gifford RH, Spahr AJ, McKarns SA. The benefits of combining acoustic and electric stimulation for the recognition of speech, voice and melodies. Audiol Neurootol. 2008;13(2):105-12. doi: 10.1159/000111782. Epub 2007 Nov 29. PMID 18057874
- [Background] Gantz BJ, Turner C, Gfeller KE. Acoustic plus electric speech processing: preliminary results of a multicenter clinical trial of the Iowa/Nucleus Hybrid implant. Audiol Neurootol. 2006;11 Suppl 1:63-8. doi: 10.1159/000095616. Epub 2006 Oct 6. PMID 17063013
- [Background] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- [Background] Gifford RH, Dorman MF, McKarns SA, Spahr AJ. Combined electric and contralateral acoustic hearing: word and sentence recognition with bimodal hearing. J Speech Lang Hear Res. 2007 Aug;50(4):835-43. doi: 10.1044/1092-4388(2007/058). PMID 17675589
- [Background] Gifford RH, Dorman MF, Shallop JK, Sydlowski SA. Evidence for the expansion of adult cochlear implant candidacy. Ear Hear. 2010 Apr;31(2):186-94. doi: 10.1097/AUD.0b013e3181c6b831. PMID 20071994
- [Background] Gifford RH, Dorman MF, Skarzynski H, Lorens A, Polak M, Driscoll CL, Roland P, Buchman CA. Cochlear implantation with hearing preservation yields significant benefit for speech recognition in complex listening environments. Ear Hear. 2013 Jul-Aug;34(4):413-25. doi: 10.1097/AUD.0b013e31827e8163. PMID 23446225
- [Background] Gifford RH, Shallop JK, Peterson AM. Speech recognition materials and ceiling effects: considerations for cochlear implant programs. Audiol Neurootol. 2008;13(3):193-205. doi: 10.1159/000113510. Epub 2008 Jan 22. PMID 18212519
- [Background] Nilsson M, Soli SD, Sullivan JA. Development of the Hearing in Noise Test for the measurement of speech reception thresholds in quiet and in noise. J Acoust Soc Am. 1994 Feb;95(2):1085-99. doi: 10.1121/1.408469. PMID 8132902
- [Background] PETERSON GE, LEHISTE I. Revised CNC lists for auditory tests. J Speech Hear Disord. 1962 Feb;27:62-70. doi: 10.1044/jshd.2701.62. No abstract available. PMID 14485785
- [Background] Skarzynski H, van de Heyning P, Agrawal S, Arauz SL, Atlas M, Baumgartner W, Caversaccio M, de Bodt M, Gavilan J, Godey B, Green K, Gstoettner W, Hagen R, Han DM, Kameswaran M, Karltorp E, Kompis M, Kuzovkov V, Lassaletta L, Levevre F, Li Y, Manikoth M, Martin J, Mlynski R, Mueller J, O'Driscoll M, Parnes L, Prentiss S, Pulibalathingal S, Raine CH, Rajan G, Rajeswaran R, Rivas JA, Rivas A, Skarzynski PH, Sprinzl G, Staecker H, Stephan K, Usami S, Yanov Y, Zernotti ME, Zimmermann K, Lorens A, Mertens G. Towards a consensus on a hearing preservation classification system. Acta Otolaryngol Suppl. 2013;(564):3-13. doi: 10.3109/00016489.2013.869059. PMID 24328756
- [Background] Spahr AJ, Dorman MF, Litvak LM, Van Wie S, Gifford RH, Loizou PC, Loiselle LM, Oakes T, Cook S. Development and validation of the AzBio sentence lists. Ear Hear. 2012 Jan-Feb;33(1):112-7. doi: 10.1097/AUD.0b013e31822c2549. PMID 21829134
- [Background] Verschuur C, Hellier W, Teo C. An evaluation of hearing preservation outcomes in routine cochlear implant care: Implications for candidacy. Cochlear Implants Int. 2016 Apr;17 Suppl 1:62-5. doi: 10.1080/14670100.2016.1152007. PMID 27099115
- [Background] Vickers D, De Raeve L, Graham J. International survey of cochlear implant candidacy. Cochlear Implants Int. 2016 Apr;17 Suppl 1:36-41. doi: 10.1080/14670100.2016.1155809. PMID 27099109
- [Background] von Ilberg CA, Baumann U, Kiefer J, Tillein J, Adunka OF. Electric-acoustic stimulation of the auditory system: a review of the first decade. Audiol Neurootol. 2011;16 Suppl 2:1-30. doi: 10.1159/000327765. Epub 2011 May 24. PMID 21606646

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-arm
Started | 44
Completed | 40
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Single-arm: Single-arm, repeated-measures study design with all subjects receiving a MED-EL cochlear implant
  MED-EL SYNCHRONY/SYNCHRONY 2 (PIN) Cochlear Implant System: Subjects were implanted with the MED-EL SYNCHRONY/SYNCHRONY 2 (PIN) Cochlear Implant System with +FLEX28 or +FLEXSOFT electrode arrays. Subjects were fit with the SONNET/SONNET 2 EAS (ear-level) and/or RONDO/RONDO 2/RONDO 3 (single-unit) external audio processors.
Arm/Group | Single-arm
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  Canada | 12
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Correct on Word Recognition in Quiet in Implanted Ear
Description: CNC (Consonant Nucleus Consonant) word scores will be calculated as percent correct at baseline and at 6 months post-activation and reported as mean percentage-point improvement at 6 months post-activation compared to baseline.
Time Frame: 6 months post-activation
Population: Analysis population includes participants in the intent-to-treat (implanted) population with 6-month data or imputed data for primary endpoint analysis.
Measure: Mean (Standard Deviation); unit: Change in percentage points
Arm/Group | Single-arm
Number analyzed (Participants) | 43
Change in percentage points | 25.6 (22.8)

2. Primary Outcome: Change in Percent Correct of Words Identified for Sentences in Noise in Implanted Ear
Description: AzBio sentence recognition in noise scores will be calculated as percent correct of words in each sentence at baseline and at 6 months post-activation and reported as mean percentage-point improvement at 6 months post-activation compared to baseline.
Time Frame: 6 months post-activation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in percentage points
Arm/Group | Single-arm
Number analyzed (Participants) | 43
Change in percentage points | 24.1 (25.3)

3. Secondary Outcome: Change in Global Score on Patient-reported Outcomes in Everyday Listening Condition
Description: APHAB (ABBREVIATED PROFILE OF HEARING AID BENEFIT) questionnaire will be used to assess subjective outcomes and reported as change in mean Global Score at 6 months post-activation compared to baseline. Letter responses from A to G on each question have a percent value, and the Global Score is an average percent value of all letters. A lower score shows less difficulty (better performance).
Time Frame: 6 months post-activation
Population: Analysis population includes participants in the intent-to-treat (implanted) population with 6-month data or imputed data for endpoint analysis. Note: not all participants completed the patient questionnaire.
Measure: Mean (Standard Deviation); unit: Change in percent, listening difficulty
Arm/Group | Single-arm
Number analyzed (Participants) | 41
Change in percent, listening difficulty | -29.5 (19.2)

4. Secondary Outcome: Number of Participants Experiencing an Adverse Device Effect (ADE)
Description: Adverse device effects will be collected for all participants through study completion and reported as the number of participants experiencing an ADE.
Time Frame: Through study completion, or at least 1 year, 4 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 44
Participants | 31

5. Secondary Outcome: Number of Participants With Residual Low-frequency Hearing
Description: HEARRING scale will be used to calculate the percent of hearing preservation for each subject by comparing average hearing thresholds from 125 to 1000 Hz at 6 months post-activation to the average at baseline.
Time Frame: 6 months post-activation
Population: Analysis population includes participants in the intent-to-treat (implanted) population with 6-month data or imputed data for endpoint analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 43
Participants
  Complete Hearing Preservation (>75%) | 3
  Partial Hearing Preservation (25-75%) | 24
  Minimal Hearing Preservation (<25%) | 4
  No Hearing Preservation | 12

6. Secondary Outcome: Change in Overall Score on Patient-reported Outcomes in Everyday Listening Condition
Description: The SSQ (Spatial and Qualities of Hearing) questionnaire will be used to assess subjective outcomes and reported as change in mean Overall Score at 6 months post-activation compared to baseline. SSQ is scored on a 10-point Likert scale where 10 shows better listening skills/experiences than 0.
Time Frame: 6 months post-activation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Single-arm
Number analyzed (Participants) | 41
Units on a scale | 1.9 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse device effects were collected through study completion for all participants. Timeframe for adverse event reporting ranged from 1 year, 4 months for the last implanted subject to 4 years, 10 months for the first implanted subject.
Arm/Group | Single-arm
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 21/44
Other Adverse Events (participants affected / at risk) | 10/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm (N=44)
Loss of residual hearing (Ear and labyrinth disorders) | 21 (21) — Loss of residual hearing after implantation
Vertigo (Ear and labyrinth disorders) | 1 (1) — Hospitalization for vertigo
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm (N=44)
Temporary loss of residual hearing (Ear and labyrinth disorders) | 7 (7) — Temporary shift in hearing thresholds improving by the study endpoint
Dizziness, imbalance, vertigo (Ear and labyrinth disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03236909/Prot_SAP_000.pdf